CLINICAL TRIAL: NCT04386850
Title: Preventive and Therapeutic Effects of Oral 25-hydroxyvitamin D3 on Coronavirus (COVID-19) in Adults
Brief Title: Oral 25-hydroxyvitamin D3 and COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRCT2020-0401046909N2; IRCT20200401046909N1 (Registry Identifier: IRCT); IRCT2020-0401046909N2 (Registry Identifier: IRCT)
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: COVID 19
Keywords: COVID 19; Vitamin D; 25-hydroxyvitamin D3; 1,25-dihydroxyvitamin D3; Viral infection; Cytokine storm; supplementation; Clinical Trial; Health Care provider; Prevention; Treatment
MeSH Terms: conditions — COVID-19; Virus Diseases; Cytokine Release Syndrome | interventions — Calcifediol

STUDY DESIGN:
Intervention Model Description: This is a multicenter randomized double-blinded placebo-controlled clinical trial with parallel groups and allocation 1:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects in a stratified random sampling method based on age, sex, BMI and serum level of 25(OH)D (<10 ng/dL vs 10 to <20 ng/dL) with serum calcium <=10.6 mg/dL will be recruited in the 25(OH)D3 or placebo group. The clinical coordinator will determine this with a computer-generated randomization program. Subjects in the case group will receive 25 mcg of 25(OH)D3 once daily at bedtime for 2 months and the control group will receive placebo daily for 2 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Infected patients with acute respiratory tract infection symptoms (e.g. fever, cough, dyspnea) with no other etiology that fully explains the clinical presentation accompanied by chest computed tomography (CT) scan findings compatible with Covid-19 or with a COVID-19 positive test by the polymerase chain reaction (PCR)
  Interventions: Drug: Oral 25-Hydroxyvitamin D3
- Prevention (Experimental): This arm of study includes the health care providers and hospital workers with a negative test for COVID-19 and a close patient relative with a negative test for COVID-19 who lives with the infected patients.
  Interventions: Drug: Oral 25-Hydroxyvitamin D3

INTERVENTIONS:
Drug: Oral 25-Hydroxyvitamin D3 — Subjects in the case group will receive 25 mcg of 25(OH)D3 once daily at bedtime for 2 months and the control group will receive placebo daily for 2 months.

SUMMARY:
The goal of this clinical trial is to investigate the therapeutic efficacy of rapidly correcting vitamin D deficiency in adults with the use of 25-hydroxyvitamin D3 [25(OH)D3] for reducing the risk of acquiring the SARS-CoV-2 (COVID-19) viral infection and mitigating morbidity and mortality associated with this infection. This evidence-based hypothesis is related to several observations. Macrophages, activated T and B lymphocytes have a vitamin D receptor and 1,25-dihydroxyvitamin D3 induces defensin protein synthesis, influences immunoglobulin production and modulates T-cell cytokine production and functions. 1,25-dihydroxyvitamin D3 also reduces the angiotensin-converting enzyme 2 (ACE2) that is believed to serve as the binding site and gateway for COVID-19 to become infectious. This is a multicenter randomized3 doubleblinded placebo-controlled study aimed at determining the benefits of 25(OH)D3 treatment for the prevention of COVID-19 infection and improving clinical outcomes in infected patients. The investigators plan to recruit 1500 subjects in 3 study groups that include hospital health providers, patients with a positive test for COVID-19 and their relatives with a negative test. Eligible subjects in each study group with a documented serum level of 25(OH)D < 20 ng/mL will be randomized. Recruited subjects will be given 25 mcg of 25(OH)D3 daily or an identically appearing placebo at the time of randomization for two months. Three hospitals will participate and the sample size is foreseen to be equally distributed between the three. Since the clinical trial is designed as minimal risk a formal committee for data monitoring is not foreseen. However, potential toxicity will be monitored every 4 weeks with a serum calcium, albumin and creatinine by the PI and the study coordinators. If the corrected serum calcium increases above 10.6 mg/dl and a repeat confirms that the calcium is above 10.6 mg/dL the subject will be dropped from the study and referred to his or her PCP. Early signs and symptoms of vitamin D toxicity associated with hypercalcemia are increased thirst, increase in frequency of urination, especially at night. The subjects will be followed up weekly by phone to ask about their sign and symptoms.

DETAILED DESCRIPTION:
Improvement in the vitamin D status i.e. total serum 25-hydroxyvitamin D in children and adults has been associated with reduced risk of upper respiratory tract infections including influenza A infection. The rationale for giving 25(OH)D3 rather than vitamin D3 is to rapidly improve the vitamin D status of the subjects who are at high risk of acquiring COVID 19 or who are infected by this very aggressive viral infection. It takes approximately 6-8 weeks to achieve a steady state blood level of 25(OH)D when ingesting a daily dose of vitamin D3 whereas ingesting 25(OH)D3 results in a rapid rise in its blood level reaching steady state within 48 hours. Based on the available literature it is reasonable to consider the possibility that vitamin D deficiency could increase risk of acquiring COVID 19 infection and exacerbating its infectivity and the body's cytokine response to it. It therefore seems plausible that the rapid improvement in vitamin D status by providing 25(OH)D3 may contribute to reducing the severity of illness caused by COVID-19, particularly in settings where hypovitaminosis D is frequent especially in people of color. Arguably, there is little evidence to date that improving the vitamin D status will reduce the infectivity risk or mitigate the devastating health consequences of COVID-19 infection. The proposed study to rapidly improve vitamin D status in adults who are at high risk of acquiring COVID- 19 or who are at risk for its morbidity and mortality will test the veracity of this evidence based hypothesis. Results from this study, especially if positive, would have far reaching global health consequences. Vitamin D3, vitamin D2 and 25-hydroxyvitamin D3 are readily available worldwide and could be quickly instituted as a rapid cost-effective method to help combat this pandemic.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old and younger than 75 years old for all study groups.
2. Meet the diagnostic criteria of COVID-19 for different types (including ordinary type, heavy type and critical type) in infected patients.
3. No medications or disorders that would affect vitamin D metabolism
4. Women must be on birth control and not pregnant
5. Ability and willingness to give informed consent and comply with protocol requirements

Exclusion Criteria:

1. Ongoing treatment with pharmacologic doses of vitamin D, vitamin D metabolites or analogues
2. Pregnant or lactating women;
3. Severe underlying diseases, such as advanced malignant tumors, endstage lung disease, etc.
4. History of elevated serum calcium >10.6 mg/dl; that is corrected for albumin concentration or subjects with a history of hypercalciuria and kidney stones.
5. Chronic hepatic dysfunction, chronic kidney disease or intestinal malabsorption syndromes including inflammatory bowel disease.
6. Supplementation with over the counter formulations of vitamin D2 or vitamin D3
7. Use of tanning bed or artificial UV exposure within the last two weeks.
8. Consuming medication affecting vitamin D metabolism or absorption (anticonvulsants, anti-tuberculosis medication glucocorticoids, HIV medications and cholestyramine).
9. Subjects with a history of an adverse reaction to orally administered vitamin D, vitamin D metabolites or analogues.
10. Subjects with a history of conditions that can lead to high serum calcium levels such as sarcoidosis, tuberculosis and some lymphomas associated with activated macrophages which increase the production of 1,25(OH)2D.
11. Inability to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
COVID-19 (SARA-Cov-2) infection | 60 days
  Percentage of patients with acute respiratory tract infection symptoms (e.g. fever, cough, dyspnea) with no other etiology that fully explains the clinical presentation accompanied by chest computed tomography (CT) scan findings compatible with Covid-19 or patients with a COVID-19 positive test by the polymerase chain reaction (PCR)
Severity of COVID-19 (SARA-Cov-2) infection | 60 days
  Percentage of mild, moderate and sever forms of COVID-19 based on WHO criteria
Hospitalization | 60 days
  Percentage of patients who need to be hospitalized
Disease duration | 60 days
  Days from the first symptom/positive test to discharge from hospital/negative test
Death | 60 days
  Rate of death due to COVID-19 during the study
Oxygen support | 60 days
  Percentage of COVID patients who need oxygen support

SECONDARY OUTCOMES:
Type of oxygen support | 60 days
  Percentage of COVID patients who require each: Nasal cannula, Non-invasive ventilation or high-flow nasal cannula, Invasive mechanical ventilation, Invasive mechanical ventilation and ECMO
Symptoms of COVID-19 | 60 days
  Percentage of COVID patients who display each: fever, dry cough, coughing sputum or blood, sore throat, headache, diarrhea and shortness of breath
Serum Levels of 25-hydroxyvitamin D3 | 60 days
  Serum Levels of 25-hydroxyvitamin D3 (ng/ml) by HPLC
Serum levels of calcium | 60 days
  Serum calcium concentration (mg/dl)
Serum levels of phosphorus | 60 days
  Serum phosphorus concentration (mg/dl)
Serum levels of creatinine | 60 days
  Serum creatinine concentration (mg/dl)
Serum levels of albumin | 60 days
  Serum albumin concentration (g/dl)
Serum levels of the blood urea nitrogen (BUN) | 60 days
  Serum concentration of the blood urea nitrogen (mg/dl)
Serum levels of the parathyroid hormone (PTH) | 60 days
  Serum concentration of the parathyroid hormone (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamadali Sahraian, MD, Study Chair — Tehran University of Medical Sciences; zhila Maghbooli, PhD, Principal Investigator — Tehran University of Medical Sciences; Michael F Holick, PhD,MD, Principal Investigator — Boston University; Arash Shirvani, MD, PhD, Principal Investigator — Boston University
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and analyzed during the current study will be available from the Study Principal Investigators (zhilayas@gmeil.com) on reasonable request .
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 9 month and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by the current study principal investigators.

REFERENCES:
- [Derived] Shakoor H, Feehan J, Al Dhaheri AS, Cheikh Ismail L, Ali HI, Alhebshi SH, Apostolopoulos V, Stojanovska L. Role of vitamin D supplementation in aging patients with COVID-19. Maturitas. 2021 Oct;152:63-65. doi: 10.1016/j.maturitas.2021.03.006. Epub 2021 Mar 16. No abstract available. PMID 33757717